CLINICAL TRIAL: NCT01539915
Title: A Single Center, Open Label Exploratory Study to Evaluate the Pharmacokinetics and Pharmacodynamics of Topically Administered BCT194 in Dermal Interstitial Fluid in Psoriatic Patients Using Open Flow Microperfusion
Brief Title: Pharmacokinetics and Pharmacodynamics of BCT194 in Psoriatic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group
Other Study IDs: CBCT194A2102; 2006-004690-10 (EudraCT Number)
Record Dates: First submitted 2012-02-22; First posted 2012-02-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Psoriasis
Keywords: Psoriasis; Stable plaque psoriasis; lesions; TNF-alpha; BCT194
MeSH Terms: conditions — Psoriasis

ARMS (1):
- BCT194 (Experimental)
  Interventions: Drug: BCT194

INTERVENTIONS:
Drug: BCT194 — Topically applied BCT194 cream (0.5%)

SUMMARY:
This study will evaluate the pharmacokinetics and pharmacodynamics of BCT194 in psoriatic patients to better understand the skin penetration of topically applied BCT194.

ELIGIBILITY:
Inclusion criteria:

* Male patients and post menopausal or surgically sterile female patients aged 18 - 75 years.
* Diagnosis of stable plaque psoriasis (with or without arthritis); diagnosed or history of psoriasis for at least 6 months prior to screening
* Psoriatic plaques accessible for microperfusion at body sites (e.g. trunk) convenient for the patients.

Exclusion criteria:

* Currently have any of the nonplaque forms of psoriasis: erythrodermic, guttate, or pustular.
* Currently have drug-induced psoriasis (new onset or exacerbation of psoriasis from beta blockers, calcium channel blockers, or lithium).
* Recent previous treatment with anti-TNF-α therapy (or other biological therapy), immunosuppressive agents such as cyclosporine, mycophenolate, pimecrolimus, or tacrolimus.
* Current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, psychiatric, or other disease which would make the patient unsuitable for the trial.
* Presence of major chronic inflammatory autoimmune diseases like rheumatoid arthritis, spondyloarthropathy, inflammatory bowel disease or systemic lupus erythematosus.
* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-04; Primary Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
change in Maximum dermal interstitial concentration of BCT194 | Day 1 and day 8
  Interstitial fluid will be collected and concentrations of BCT194 determined determined on Day 1 and Day 8 at several timepoints
Area under the curve interstitial concentrations of BCT194 | day 1 and day 8
  Interstitial fluid will be collected and concentrations of BCT194 determined on Day 1 and Day 8 at several timepoints

SECONDARY OUTCOMES:
Concentrations of locally produced tumor necrosis factor-alpha (TNF-alpha) | day 1 and day 8
  Interstitial fluid will be collected and concentrations of Tumor Necrosis Factor alpha determined determined on Day 1 and Day 8 at several timepoints
Change in plaque PASI scores of psoriasis lesions | day 1 and day 8
  Treatment areas will be assessed clinically at baseline and Day 8
BCT194 concentrations in skin biopsies | day 1 and day 8
  Biopsies of lesional and nonlesional skin will be collected 4 hours post dose on Day 1 and Day 8 for measurement of BCT194 concentration.
Change in Local tolerability score | Pre-dose, Day 1, Day 2, Day 3, Day 5, Day 8, Day 9 and Day 13
  Local tolerability assessed using a validated score (0-4) for each treatment area
  Safety Issue: Treatment sites will be visually assessed for visible reaction to the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis Investigative Site, Graz, Austria